CLINICAL TRIAL: NCT05483855
Title: Telehealth-delivered HealthcaRe to ImproVe Care (THRIVE) as an Integral Component of Remote Therapeutic Monitoring (RTM)
Brief Title: Telehealth-delivered HealthcaRe to ImproVe Care
Acronym: THRIVE
Status: Recruiting | Type: Observational
Sponsor: Attune Health Research, Inc. (Industry)
Collaborators: Rheumatology Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: THRIVERTM
Record Dates: First submitted 2022-07-27; First posted 2022-08-02 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Telemedicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Objective 1: Telehealth Visit: Any rheumatology patient, seen and treated by a participating physician, who is 19 years and older, with the target condition(s) of interest, and is already scheduled for a telehealth visit.
  Interventions: Other: Objective 1 Only: Telehealth Satisfaction Survey
- Objective 2: ArthritisPower App: Patients diagnosed with Rheumatoid Arthritis who already have a pre-scheduled in-office visit.
  Interventions: Other: Objective 2 Only: ArthritisPower Joint Assessment

INTERVENTIONS:
Other: Objective 1 Only: Telehealth Satisfaction Survey — Participants must complete a telehealth satisfaction survey rating their standard of care telehealth visit on a scale of 1 to 10, with 1 denoting low satisfaction and 10 denoting high satisfaction.
  Groups: Objective 1: Telehealth Visit
Other: Objective 2 Only: ArthritisPower Joint Assessment — RA patients must complete a self-assessment examination of their joints using the ArthritisPower app prior to their in-office visit, where a repeat joint assessment is performed by participating physician.
  Groups: Objective 2: ArthritisPower App

SUMMARY:
Objective 1:

Evaluate patients' satisfaction with their telehealth care and determine factors associated with satisfaction.

Objective 2:

Deploy PROs and patient self-assessment tools, specifically a patient-facing instructional in-app tool that instructs RA patients how to perform self-assessment examinations to observe and report the number of tender and swollen joint counts.

DETAILED DESCRIPTION:
Objective 1:

Any rheumatology patients, seen and treated by participating physicians, who are 19 years and older with the target condition(s) of interest and are pre-scheduled for a telehealth visit, are eligible to participate and will be invited. The desired enrollment target is 1500 respondents shared amongst the 12 participating rheumatologists. One week before the scheduled telehealth visit, patients who have agreed to participate will receive electronic communication from participating physicians' offices notifying them that they will be asked to complete a survey about their satisfaction with their telehealth visit after its conclusion. Within approximately 1 business day following the standard of care telehealth visit, participants will be sent a text via an Electronic Data Capture system inviting them to participate in the survey. Upon clicking on the survey link provided in the text message, participants will be prompted to rate their level of satisfaction with their telehealth visit on a scale of 1 to 10, with a score of 1 denoting low satisfaction and a score of 10 denoting high satisfaction. Selection of a score of 8 or lower will prompt participants to answer additional subsequent questions that queries them to explain the reasons for their unsatisfactory patient experience. Data from the surveys will be linked back to participants; electronic health record data to evaluate characteristics such as age, health conditions, disease activity, treatments, social determinants of health, multi-morbidity, PROs, medicated based multi-morbidity, driving distance from a patient's home to the physician's office, rural/urban status, disease indication for the telehealth visit associated with the unsatisfactory telehealth encounter. Data from participant surveys will be linked with Electronic Health Record (EHR) data to analyze factors associated with satisfaction. Logistic regression with generalized estimating equations (GEE) will be used to model factors associated with low telehealth satisfaction, controlling for site clustering.

Objective 2:

8-10 patients with Rheumatoid Arthritis from each site of the same 12 participating physicians who have already-scheduled in-office visits will be invited to participate. The target recruitment goal is approximately 100 patients, which, after accounting for attrition would allow for an analytic sample of about 70-80 Rheumatoid Arthritis patients. Patients will be recruited via in-person solicitation, email, patient portal, text-messaging, or a combination of these. Interested patients will be sent a link by email or text message to join the ArthritisPower registry after which a unique and custom generated password will be generated that has no relationship to identifying patient information. After registration, participants will be prompted to complete the in-app instructional tool for self-assessment examination of their joints in addition to several RA-related patient reported outcomes. The assessment in ArthritisPower must be completed as soon as participant has received the link to register for the application. Within 3 business days of the ArthritisPower self-assessment, participants will have their scheduled in-office examination of their joints by their physician to collect the provider joint examination findings and other physician data in an EDC system. If there has been more than a 7-business day gap between the patient self-assessment in the ArthritisPower app, and the in-person exam, that patient will be ineligible for analysis and will be replaced. The correlation between patient joint count will be analyzed. The investigators will examine and compare the patient and rheumatology provider's render and swollen joint count summed scores and Perason and Spearman's correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* Must be 19 years or older.
* Must have a prior diagnosis of Rheumatoid Arthritis.
* Must be able to read and write in English or Spanish.

Exclusion Criteria:

* Younger than 19 years of age
* Does not have a prior diagnosis of Rheumatoid Arthritis.
* Unable to read and write in English or Spanish

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Rheumatoid Arthritis seen in a Rheumatology Clinic.
Sampling Method: Probability Sample
Enrollment: 1580 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Correlation between patient joint count and provider joint count | Immediately after the intervention
  The investigators will examine and compare the patient and rheumatology provider's tender and swollen joint count summed scores and Pearson and Spearman's correlation coefficient (if the data is non-normally distributed). The investigators will also calculate a typical Clinical Disease Index (CDAI) for RA which is a composite score of TJC28 + SJC28 + Patient Global + Provider Global and correlate with the patient [p] CDAI ([p]TJC28 + [p]SJC28 + Patient Global + Provider Global). Disease remission for RA is denoted by a CDAI composite score of less than or equal to 2.8 while high RA disease activity is denoted by a CDAI score of 22 or greater. The investigators will also compute weighted kappa statistics, comparing the 4x4 table of remission, low moderate, and high disease activity categories, using the traditional CDAI cut points (2.8, 10, and 22).

CONTACTS AND LOCATIONS:
Locations (1):
- Attune Health Research Inc, Beverly Hills, California, United States